CLINICAL TRIAL: NCT02804438
Title: Establishing Normative Data for Pupillometer Assessments in Neuro-Intensive Care
Acronym: ENDPANIC
Status: Recruiting | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: NeurOptics Inc. (Industry)
Responsible Party: Principal Investigator, DaiWai Olson, Professor, University of Texas Southwestern Medical Center
Other Study IDs: STU 062015-005
Record Dates: First submitted 2016-05-03; First posted 2016-06-17 (Estimated); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Critical Illness; Neuropathy
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to collect a large amount of data that may assist in addressing the gap in knowledge of understanding pupillometer readings using a pupillometer device.

The aim of this project is to establish normative values for pupillometer data. Measures of central tendency will be developed for the variables provided by automated pupillary exams, which will provide an enhanced understanding of clinically appropriate pupil values for size, reactivity, and neurological pupil index.

DETAILED DESCRIPTION:
Data will be collected on patients in the intensive care units at the selected hospitals on patients who have been assigned, by the attending physician, to have regular pupillary assessments, and in whom staff nurses are performing pupillary assessments with the pupillometer. While a sample size estimate would be considered inappropriate for registry development, power analysis techniques were used to examine the potential of this registry to generate adequate information to begin to fully describe normative data for pupillary exams. Using the assumption that the desire is to understand neurological pupil index (NPi) and size differences within 0.1, and that the spread of data would be approximately normally distributed, a minimum of 3,250 observations is required (alpha = 0.05, beta = 0.80). It must, however, be repeated that this is simply a rough estimate. The registry data generated will, in fact, be the source of data from which future studies will be powered.

ELIGIBILITY:
Inclusion Criteria:

* Data will be collected on patients admitted to enrolling hospitals who have been assigned, by the attending physician, to have regular pupillary assessments, and in whom staff nurses are performing pupillary assessments with the pupillometer.

Exclusion Criteria:

* Out-patients
* Patients that do not have orders for regular pupillary assessments

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: In-patient
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-07 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Oculomotor evaluation of pupillary variance during ICU admission | Daily at 9:00am
  Pupil size and reactivity per neurological pupil index

CONTACTS AND LOCATIONS:
Locations (1):
- Maria E Denbow, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Privitera CM, Neerukonda SV, Aiyagari V, Yokobori S, Puccio AM, Schneider NJ, Stutzman SE, Olson DM; END PANIC Investigators. A differential of the left eye and right eye neurological pupil index is associated with discharge modified Rankin scores in neurologically injured patients. BMC Neurol. 2022 Jul 22;22(1):273. doi: 10.1186/s12883-022-02801-3. PMID 35869429
- [Derived] Campos YA, Rana P, Reyes RG, Mazhar K, Stutzman SE, Atem F, Olson DM, Aiyagari V. Relationship Between Automated Pupillometry Measurements and Ventricular Volume in Patients With Aneurysmal Subarachnoid Hemorrhage. J Neurosci Nurs. 2022 Aug 1;54(4):166-170. doi: 10.1097/JNN.0000000000000657. Epub 2022 Jun 21. PMID 35776519
- [Derived] Thakur B, Nadim H, Atem F, Stutzman SE, Olson DM. Dilation velocity is associated with Glasgow Coma Scale scores in patients with brain injury. Brain Inj. 2021 Jan 5;35(1):114-118. doi: 10.1080/02699052.2020.1861481. Epub 2020 Dec 21. PMID 33347373